CLINICAL TRIAL: NCT06112704
Title: A Phase 2, Open-label, Multi-center Study to Evaluate the Efficacy, Safety, Pharmacokinetics and Immunogenicity of HS-20093 in Patients with Advanced Esophageal Carcinoma and Other Advanced Solid Tumors (ARTEMIS-005)
Brief Title: HS-20093 in Patients with Advanced Esophageal Carcinoma and Other Advanced Solid Tumors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hansoh BioMedical R&D Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HS-20093-203
Record Dates: First submitted 2023-10-29; First posted 2023-11-01 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Advanced Solid Tumor
Keywords: Advanced solid tumor; Esophageal Carcinoma; B7-H3; antibody-drug conjugate (ADC); HS-20093
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Phase IIa: Cohort 1 (Experimental): Participants with advanced esophageal squamous cell carcinoma will be administered HS-20093.
  Interventions: Drug: HS-20093
- Phase IIa: Cohort 2 (Experimental): Participants with advanced esophageal adenocarcinoma and gastroesophageal junction adenocarcinoma will be administered HS-20093.
  Interventions: Drug: HS-20093
- Phase IIa: Cohort 3 (Experimental): Participants with other advanced solid tumor will be administered HS-20093.
  Interventions: Drug: HS-20093
- Phase IIb (Experimental): Participants with advanced esophageal squamous cell carcinoma will be administered HS-20093.
  Interventions: Drug: HS-20093

INTERVENTIONS:
Drug: HS-20093 — Intravenous (IV) infusion of HS-20093 Q3W; Participants will receive continuous treatment until the end of the study in the absence of unacceptable toxicities and confirmed disease progression.

SUMMARY:
HS-20093 is a humanized IgG1 antibody-drug conjugate (ADC) which specifically binds to B7-H3, a target wildly expressed on solid tumor cells. The objectives of this study are to investigate the anti-tumor activity, safety, pharmacokinetics and immunogenicity of HS-20093 in Chinese advanced esophageal carcinoma and other solid tumor patients.

DETAILED DESCRIPTION:
This is an open-label, multi-center phase 2 study in Chinese adult participants with recurrent, locally advanced or metastatic esophageal carcinoma or other advanced solid tumors, which is designed to investigate the efficacy, safety, pharmacokinetics and immunogenicity of HS-20093. This study will consist of two parts: phase IIa and phase IIb.

Part 1 (phase IIa) will conducted in participants with relapsed, locally advanced or metastatic esophageal carcinoma and other advanced solid tumor. Subjects will receive one dose levels of HS-20093 intravenously every 3 weeks.

Part 2 (phase IIb) will enroll participants with relapsed, locally advanced or metastatic esophageal squamous cell carcinoma. One dose levels of HS-20093 will be administered as an intravenous (IV) infusion every 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women aged more than or equal to (≥) 18 years.
2. Histologically or cytologically confirmed, relapsed, locally advanced or metastatic esophageal carcinomas and other advanced solid tumor.
3. At least one extra measurable lesion according to RECIST 1.1 (cavity structures such as oesophagus cannot serve as measurable lesions).
4. Agree to provide fresh or archival tumor tissue and blood samples.
5. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0~1.
6. Estimated life expectancy >12 weeks.
7. Agree to use medically accepted methods of contraception.
8. Men or women should be using adequate contraceptive measures throughout the study.
9. Females subjects must not be pregnant at screening or have evidence of non-childbearing potential.
10. Signed and dated Informed Consent Form.

Exclusion Criteria:

Any of the following would exclude the subject from participation in the study:

1. Treatment with any of the following:

   Previous or current treatment with B7-H3 targeted therapy Any cytotoxic chemotherapy, investigational agents and anticancer drugs within 14 days prior to the first scheduled dose of HS-20093 Prior treatment with a monoclonal antibody within 28 days prior to the first scheduled dose of HS-20093 Local radiotherapy for palliation within 2 weeks of the first dose of study drug, or patients received more than 30% of the bone marrow irradiation, or large-scale radiotherapy within 4 weeks prior to the first scheduled dose of HS-20093 Major surgery within 4 weeks prior to the first scheduled dose of HS-20093
2. Subjects with previous or concurrent malignancies
3. Significant tumor invasion into adjacent organs (aorta or trachea) of esophageal lesions leading to higher risk of bleeding or fistula
4. Inadequate bone marrow reserve or organ dysfunction.
5. Evidence of cardiovascular risk
6. Evidence of current severe or uncontrolled systemic diseases
7. Evidence of mucosal or internal bleeding within 1 month prior to the first scheduled dose of HS-20093
8. Severe infections occured within 4 weeks before the first dose
9. The presence of active infectious diseases has been known before first dose such as hepatitis B, hepatitis C, ect
10. History of neuropathy or mental disorders
11. Pregnant or lactating female
12. History of severe hypersensitivity reaction, severe infusion reaction or idiosyncrasy to drugs chemically related to HS-20093 or any of the components of HS-20093
13. Known vaccination or hypersensitivity of any level within 4 weeks prior to the first scheduled dose of HS-20093
14. Unlikely to comply with study procedures, restrictions, and requirements in the opinion of the investigator
15. Any disease or condition that, in the opinion of the investigator, would compromise subject safety or interfere with study assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2024-02-06 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) determined by investigators according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. | From the first dose up to disease progression（PD）or withdrawal from study，whichever comes first，assessed up to 24 months.
  ORR was defined as the percentage of participants who achieved a best overall response (BOR) of confirmed Complete Response (CR) or Partial Response (PR), assessed by investigators based on RECIST version 1.1[Confirmed CR/PR assessment require at least one repeat (≥4 weeks)].

SECONDARY OUTCOMES:
DOR assessed by RECIST 1.1 criteria | From the first dose up to PD or death, whichever came first, assessed up to 24 months.
  DOR was defined as the period from the first occurrence of CR or PR to PD or death from any cause. If no PD or death after CR/PR, the cut-off date of progression-free survival (PFS) would be used [Confirmed CR/PR assessment require at least one repeat (≥4 weeks)
Disease Control Rate (DCR) assessed by RECIST 1.1 criteria | From the first dose up to PD or withdrawal from study, whichever came first, assessed up to 24 months.
  DCR was evaluated by the number of participants with best overall response of CR, PR and stable disease (SD) [Confirmed CR/PR assessment require at least one repeat (≥4 weeks); SD shall be assessed at least 5 weeks after the first dose.
PFS assessed by RECIST 1.1 criteria | From the first dose up to PD or death，whichever came first, assessed up to 24 months.
  PFS was defined as the time from first dose or random assignment (if any) to PD or death from any cause
Overall survival (OS) | From the first dose up to PD or death，whichever came first, assessed up to 24 months.
  OS was defined as the time from the first dose or random assignment (if any) to death from any cause
Incidence and severity of adverse events | From the first dose until 90 days after the last dose
  AE assessed by investigator exclusively related to subject's underlying disease or medical condition [graded according to the NCI Common Terminology Criteria for Adverse Events (CTCAE), Version 5.0]. Any untoward medical occurrence in a clinical study participant, whether or not considered related to the medicinal product. Incidence and severity of AEs are assessed according to vital signs, laboratory variables, physical examination, electrocardiogram, etc
Characterize the pharmacokinetic parameters of HS-20093 | Cycle 1 Day 1 up to 90 days after the last dose
  Characterize the pharmacokinetic parameters of HS-20093
Assess the incidence of anti-drug antibodies (ADAs) | Cycle 1 Day 1 up to 90 days after the last dose
  Serum samples were collected for the determination of anti-drug antibody (ADA) at designated time points

CONTACTS AND LOCATIONS:
Locations (21):
- China (21):
  - Anhui Provincial Cancer Hospital, Hefei, Anhui
  - Fujian Provincial Tumor Hospital, Fujian, Fujian
  - The 900th Hospital of the Joint Service Support Force of the Chinese People's Liberation Army, Fuzhou, Fujian
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Tumour Hospital of Anyang city, Anyang, Henan
  - The First Affiliated Hospital of Henan University of Science & Technology, Luoyang, Henan
  - Nanyang Central Hospital, Nanyang, Henan
  - The First Affiliated Hospital of Xinxiang Medical University, Xinxiang, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Tongji Hospital, affiliated with Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Nantong Tumor Hospital, Nantong, Jiangsu
  - Jiangyin People's Hospital, Wuxi, Jiangsu
  - Jiangxi Provincial Tumor Hospital, Nanchang, Jiangxi
  - Liaoning Cancer Hospital, Shenyang, Liaoning
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Affiliated Hospital of Jining Medical University, Jining, Shandong
  - Sichuan Cancer Hospital&Institude, Sichuan Cancer Center,Affiliate Cancer Hospital Of University Of Electronic Science and Technology of China, Chengdu, Sichuan
  - The Affiliated Cancer Hospital of Xinjiang Medical University, Ürümqi, Xinjiang